CLINICAL TRIAL: NCT00781846
Title: A Phase I Trial of Oral Deforolimus (AP23573; MK-8669), an mTOR Inhibitor, in Combination With Bevacizumab for Patients With Advanced Cancers
Brief Title: Trial of Deforolimus in Combination With Bevacizumab for Patients With Advanced Cancers (8669-010)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-010; AP23573-08-111
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Solid Tumor
MeSH Terms: interventions — ridaforolimus; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 30mg QDx5/wk ridaforolimus plus 10mg/kg Q2wks bevacizumab for 4 weeks
  Interventions: Drug: ridaforolimus; Drug: bevacizumab
- 2 (Experimental): 40mg QDx5/wk ridaforolimus plus 10mg/kg Q2wks bevacizumab for 4 weeks
  Interventions: Drug: ridaforolimus; Drug: bevacizumab
- 3 (Experimental): 40mg QDx5/wk ridaforolimus plus 15mg/kg Q3wks bevacizumab for 3 weeks
  Interventions: Drug: ridaforolimus; Drug: bevacizumab

INTERVENTIONS:
Drug: ridaforolimus — oral tablets, daily for 5 days/week
  Other Names: deforolimus; AP23573; MK-8669; ridaforolimus was also known as deforolimus until May 2009
Drug: bevacizumab — IV infusion
  Other Names: avastin

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and recommended phase 2 dose of oral ridaforolimus administered in combination with intravenous bevacizumab in patients with advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Advanced or metastatic solid tumor malignancy
* ECOG performance status of less than or equal to 1
* Life expectancy of greater than 3 months
* At least 4 weeks must have elapsed between prior investigational therapy, chemotherapy, or radiotherapy, and the first dose of deforolimus
* Adequate hematological, hepatic and renal function
* Serum cholesterol less than or equal to 350 mg/dL and triglycerides less than or equal to 400 mg/dL
* Signed informed consent
* Women of childbearing potential must have a negative serum pregnancy test within 7 days of starting therapy and must use an approved contraceptive method from time of screening until 30 days after the last dose of study drug

Exclusion Criteria:

* Tumor location in close proximity to a major blood vessel
* History of brain metastases, spinal cord compression, or carcinomatous meningitis. Primary brain tumors (for example, glioblastoma) are allowed.
* New brain metastases, spinal cord compression, or leptomeningeal metastases on screening CT scan or MRI
* Hemoptysis or hematemesis within 28 days prior to entering the trial
* Clinical significant unexplained bleeding within 28 days prior to entering the trial
* Uncontrolled hypertension
* Proteinuria at screening
* Clinically significant cardiovascular disease
* Newly diagnosed or poorly controlled type 1 or 2 diabetes
* Active infection requiring prescribed intervention
* Other concurrent illness that, in the Investigator's judgement, would either compromise the patient's safety or interfere with the evaluation of the safety of the study drug
* Major surgery within 28 days before trial entry, or any incompletely healed surgical incision; minor surgery or procedures within 7 days
* Pregnant or breastfeeding
* Known allergy to macrolide antibiotics
* Known hypersensitivity to any component of bevacizumab
* Concurrent treatment with medications that strongly induce or inhibit cytochrome P450 (CYP3A)
* Known history of HIV sero-positivity
* Any condition in the Investigator's judgement that renders the patient unable to fully understand and provide informed consent and/or comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Identification of recommended phase 2 dose of ridaforolimus in combination with bevacizumab | Duration of the trial

SECONDARY OUTCOMES:
Characterize the overall safety and tolerability of ridaforolimus in combination with bevacizumab | Duration of the study
Description of the anti-tumor activity of ridaforolimus in combination with bevacizumab | Duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Frank Haluska, MD, PhD, Study Director — Ariad Pharmaceuticals

REFERENCES:
- [Result] Nemunaitis J, Hochster HS, Lustgarten S, Rhodes R, Ebbinghaus S, Turner CD, Dodion PF, Mita MM. A phase I trial of oral ridaforolimus (AP23573; MK-8669) in combination with bevacizumab for patients with advanced cancers. Clin Oncol (R Coll Radiol). 2013 Jun;25(6):336-42. doi: 10.1016/j.clon.2013.02.005. Epub 2013 Apr 21. PMID 23615181